CLINICAL TRIAL: NCT01645358
Title: Hypercapnic Acute Respiratory Failure: Is the Helmet an Effective Interface?"
Brief Title: Helmet Ventilation in Acute Hypercapnic Respiratory Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, Chief Respiratory and Critical care, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1222
Record Dates: First submitted 2012-03-22; First posted 2012-07-20 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Hypercapnic Respiratory Failure; Chronic Obstructive Pulmonary Disease
Keywords: COPD; NIV; Acute Hypercapnic Respiratory Failure; COPD patients with hypercapnic respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency; Pulmonary Disease, Chronic Obstructive | interventions — Head Protective Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Helmet to deliver NIV (Experimental)
  Interventions: Device: Helmet (Starmed)
- Total Face to deliver NIV (Active Comparator)
  Interventions: Device: Total Face mask (Respironics)

INTERVENTIONS:
Device: Helmet (Starmed) — The helmet is a kind of interface similar to a hood to deliver NIV
  Other Names: Starmed Helmet
  Arms: Helmet to deliver NIV
Device: Total Face mask (Respironics) — The total face mask is the "classical" interface for NIV delivery
  Other Names: Respironics Performax or similar
  Arms: Total Face to deliver NIV

SUMMARY:
Lack of tolerance to the treatment, makes the interface choice for non-invasive ventilation (NIV) one of the key factor. To date the helmet is rarely used in Acute Hypercapnic Respiratory Failure (AHRF), because of its large dead space, despite in hypoxic respiratory failure, it is largely employed as a "rotating" strategy when the facial mask is poorly tolerated.

In a multicenter randomized controlled trial, the investigators will compare the clinical efficacy of a new helmet designed to specifically improve the performance in chronic obstructive pulmonary disease (COPD) versus a full face mask during an episode of AHRF.

ELIGIBILITY:
Inclusion Criteria:

* pH < 7,35 and PaCO2 > 45 mmHg
* respiratory rate > 20 b/min

Exclusion Criteria:

* hypoxic respiratory failure
* coma
* inability to stand NIV
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Arterial Blood gases | at 1 hour after the start of NIV

SECONDARY OUTCOMES:
Arterial Blood Gases | Once a day at 8 am until discharge

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Sant'Orsola malpighi Hospital, Bologna
  - Sant'Orsola Malpighi, Bologna

REFERENCES:
- [Derived] Pisani L, Mega C, Vaschetto R, Bellone A, Scala R, Cosentini R, Musti M, Del Forno M, Grassi M, Fasano L, Navalesi P, Nava S. Oronasal mask versus helmet in acute hypercapnic respiratory failure. Eur Respir J. 2015 Mar;45(3):691-9. doi: 10.1183/09031936.00053814. Epub 2014 Dec 10. PMID 25504992